CLINICAL TRIAL: NCT02738502
Title: An Open-label Phase II Pilot Study of Prevention of Perinatal Transmission of HIV-1 Without Nucleoside Reverse Transcriptase Inhibitors
Brief Title: Prevention of Perinatal Transmission of HIV-1 Without Nucleoside Reverse Transcriptase Inhibitors
Acronym: MONOGEST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 168 MONOGEST
Record Dates: First submitted 2016-03-23; First posted 2016-04-14 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Maternal-fetal Infection Transmission
Keywords: HIV; prevention of mother-to-child transmission; Ritonavir boosted darunavir monotherapy
MeSH Terms: interventions — Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Group (Experimental): Intervention: Darunavir monotherapy darunavir/ritonavir 600 mg/100mg twice day in monotherapy.
  Interventions: Drug: darunavir monotherapy

INTERVENTIONS:
Drug: darunavir monotherapy — darunavir 600 mg + ritonavir 100 mg 2 times 24 (DRV/r) monotherapy started after checking the tolerance of DRV/r600 mg/100 mg twice daily to replace whatever prior ARVs were used, while maintaining the NRTI backbone for 2 weeks.
  Other Names: ritonavir

SUMMARY:
The overall goal is to study the feasibility of darunavir/ritonavir (DRV/r) monotherapy as treatment simplification (switch) in pretreated pregnant women, associated with neonatal prophylaxis with nevirapine, constituting a PMTCT strategy without any Nucleoside Reverse Transcriptase Inhibitor (NRTIs) .

DETAILED DESCRIPTION:
90 participants will be enrolled and switch to darunavir monotherapy early in pregnancy (before 16 weeks of amenorrhea) in order to reduce exposure to the antiretroviral nucleos(t)ide analogues. The study treatment during the pregnancy is: darunavir 600 mg + ritonavir 100 mg 2 times 24 (DRV/r) monotherapy This regimen will be started after checking the tolerance of DRV/r 600 mg/100 mg twice daily (recommended dosage for pregnancy in French national recommendations) to replace whatever prior antiretrovirals (ARVs) were used, while maintaining the NRTI backbone for 2 weeks. Woman already receiving a triple drug combination with DRV/r will proceed directly to treatment simplification. If clinical tolerance of DRV/r is satisfactory after 2 weeks, nucleos(t)ides will be stopped. In case of intolerance, the treatment will be determined by the investigator but follow-up of the patient will continue.

No zidovudine will be administered at delivery in case of virological control, according to French Guidelines (Morlat Report 2015).

After delivery, the choice of maternal antiretrovial therapy (ART) is left to the discretion of the clinician and patient.

The mothers are followed up monthly until delivery and the last visit is planes at W4-W6 postpartum. Virological efficacy and safety will be assessed monthly.

In neonates, the prophylactic treatment, nevirapine oral solution, will be administrated as soon as possible in the first 12 hours of life and then for 14 days, once a day at a daily dose of 15 mg for a birthweight ≥ 2.5 kg ; 10 mg for a birthweight ≥ 2 kg and < 2.5 kg and 2 mg / kg for a birthweight < 2 kg (WHO Guidelines 2013 - French Guidelines, "Morlat Report" 2015).

Clinical and virological monitoring will be performed at Day 3, Day 15 in case of hospitalization, M1, M3 and M6.

Statistical Methods The analysis of the primary endpoint is the proportion of virological success (VL < 50 copies/mL at delivery among women remaining on DRV/r). All changes in antiretroviral therapy because of VL ≥ 50 copies/ml will be considered as failures. Women who change antiretroviral therapy for other reasons and/or when pregnancy outcome is before 22 weeks of amenorrhea and < 500g (non-viable pregnancy according to WHO) will be removed from the denominator.

Analysis of treatment changes, tolerance for the mother and child and factors associated with virological failure will be done by estimating percentages (categorical variables), average and median (continuous variables) with their intervals 95% confidence, overall and compared between the groups with virological success or failure per protocol (primary endpoint) or by intention to treat (secondary endpoint). The evolution of the parameters measured in children at birth, at 1, 3, and 6, months will be explored using non-parametric curves and compared between groups by repeated data taking into account the nonlinearity developments.

No interim analysis is planned.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman, under 15 weeks gestational age at screening
* Documented Human Immunodeficiency Virus (HIV) HIV-1 infection (serology and/or plasma HIV RNA viral load)
* Current treatment with at least two ARVs
* Virological suppression for at least 12 months, defined by a PVL < 50 copies / mL. A blip (transiently ≥ 50 but < 400 copies/mL) will not be considered as an exclusion criterion, if it is followed by 2 successive controls with CV < 50 at least one month before enrollment
* Plasma viral load < 50 copies/mL at pre-inclusion
* CD4 ≥ 250 cells/mm3 at pre-inclusion
* Informed written consent
* Health care coverage

Inclusion criteria for the child :

* Mother enrolled in the trial
* Informed written consent by parents or legal guardians

Exclusion Criteria:

* Infection by HIV-2
* History of treatment failure and/or resistance with any Protease Inhibitor (PI). Treatment failure is defined by a viral replication (≥ 50 copies/mL) during antiretroviral treatment. An increasing CV due to treatment interruption will not be considered as a failure, providing that the absence of resistance mutations to at least one PI can be confirmed by genotyping.
* Documented CD4 lymphocyte less than 200/mm3
* Known intolerance to darunavir or ritonavir
* Hepatitis B Virus (HBV) co-infection (HBs Ag-positive and/or detectable HBV DNA) on therapy with analogs (tenofovir, emtricitabine, lamivudine)
* Known resistance of maternal viral strain to darunavir or nevirapine
* Intended absence (travel abroad, moving ...)
* Expected delivery in a maternity hospital not participating in the trial
* Participation in the trial during previous pregnancy
* Persons under guardianship or deprived of liberty by a judicial or administrative decision

Exclusion criteria for the child:

* Refusal by parent (s) or legal guardian (s)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Success rate, defined by plasma viral load (PVL) <50 copies / mL near delivery with DRV/r monotherapy. Failure is defined as PVL > 50 copies / mL and/or change of antiretroviral therapy during pregnancy for PVL ≥ 50 copies / mL. | At delivery (around 6 months after enrollment in the study).

SECONDARY OUTCOMES:
Plasma viral load (PVL) <50 copies / mL at delivery, Intention-to-treat (ITT) analysis | At delivery (around 6 months after enrollment in the study).
Incidence of treatment changes for inefficacy, defined as PVL≥ 50 copies / mL at 2 successive controls. | Every month from Month1 up to the delivery.
Incidence of treatment changes for intolerance / toxicity. | Every month from Month1 up to the delivery.
Incidence of treatment changes for other reasons. | Every month from Month1 up to the delivery.
Factors associated with inefficacy (HIV-1 DNA). Inefficacy is defined as maternal plasma viral load > 50 copies/mL at delivery and/or change of antiretroviral therapy at any time from enrollment through delivery for plasma viral load > 50 copies/mL. | Every month from Month1 up to the delivery.
  The following quantitative variables will be compared between women with inefficacy and those with virological success (plasma viral load < 50 copies/mL under darunavir/ritonavir) : HIV-1 DNA (total HIV-DNA log10 copies/million peripheral blood mononuclear cells by the ANRS technique).
Factors associated with inefficacy (lymphocytes T CD4+ count). | Every month from Month1 up to the delivery.
  Inefficacy is defined as maternal plasma viral load > 50 copies/mL at delivery and/or change of antiretroviral therapy at any time from enrollment through delivery for plasma viral load > 50 copies/mL. The following quantitative variables will be compared between women with inefficacy and those with virological success (plasma viral load < 50 copies/mL under darunavir/ritonavir) : CD4+ lymphocyte count/microL.
Factors associated with inefficacy (CD4 nadir). Inefficacy is defined as maternal plasma viral load > 50 copies/mL at delivery and/or change of antiretroviral therapy at any time from enrollment through delivery for plasma viral load > 50 copies/mL. | Every month from Month1 up to the delivery.
  The following quantitative variables will be compared between women with inefficacy and those with virological success (plasma viral load < 50 copies/mL under darunavir/ritonavir) : CD4+ lymphocyte/microL nadir.
Factors associated with inefficacy (duration of undetectable plasma viral load before pregnancy). | Every month from Month1 up to the delivery.
  Inefficacy is defined as maternal plasma viral load > 50 copies/mL at delivery and/or change of antiretroviral therapy at any time from enrollment through delivery for plasma viral load > 50 copies/mL. The following quantitative variables will be compared between women with inefficacy and those with virological success (plasma viral load < 50 copies/mL under darunavir/ritonavir) : duration of undetectable plasma viral load before pregnancy (months).
Adverse pregnancy outcomes (preterm birth) | At delivery
  preterm birth : < 37 weeks gestational age from last menstrual period)
Adverse pregnancy outcomes (fetal loss) | Every month from Month1 up to the delivery.
  Fetal loss defined as all stillbirths and spontaneous abortions before 22 weeks gestation
Adverse pregnancy outcomes (low birth weight) | At delivery
  low birth weight < 3d percentile adjusted for gestational age and sex
Adverse pregnancy outcomes (low Apgar : < 7 at 5 minutes) | At delivery
Adverse pregnancy outcomes (congenital malformations) | At delivery
  Malformations according to the European Surveillance of Congenital Anomalies (EUROCAT) classification)
Tolerance in children (hematological examinations). | At delivery, Day 3, 15, Month1, 3 and 6
  Hemoglobin, red blood cell count, white blood cell counts and differentials and platelet counts /microL, and mean corpuscular volume in fL
Tolerance in children (biochemical examinations). | At delivery, Day 3, 15, Month1, 3 and 6
  AST and ALT, total bilirubin, lipase, sodium, potassium, urea, creatinine, calcium, phosphorus, lactates
Interruption rate of postnatal nevirapine (NVP) within 2 weeks of life and patterns; | Day 3, Day15
Any case of mother to child transmission would be considered a serious adverse event (SAE) and analyzed immediately. | Day 3, Month1, Month 3 and Month 6.

CONTACTS AND LOCATIONS:
Overall Officials: François DABIS, Pr, MD, Study Director — ANRS, Emerging Infectious Diseases
Locations (23):
- France (23):
  - CH Victor Dupouy, Argenteuil
  - Hôpital Jean Verdier, Bondy
  - Groupe hospitalier Pellegrin, Bordeaux
  - Hôpital Saint André, Bordeaux
  - Hôpital Antoine Béclère, Clamart
  - Hôpital Louis Mourier, Colombes
  - Hôpital Sud Francilien, Corbeil-Essonnes
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital de la croix Rousse, Lyon
  - Hôtel Dieu, Nantes
  - CHU Archet 1, Nice
  - Hôpital Lariboisiere, Paris
  - Hôpital Armand Trousseau, Paris
  - Hôpital la Pitié Salpétrière, Paris
  - Groupe hospitalier Cochin-Broca- Hôtel Dieu, Paris
  - HEGP, Paris
  - Hôpital Necker Enfant malades, Paris
  - Hôpital Bichat - Claude Bernard, Paris
  - Hôpital Tenon, Paris
  - CHU de Perpignan, Perpignan
  - CHU Rennes Hôpital Pontchaillou, Rennes
  - Hôpital Foch, Suresnes
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arribas JR, Girard PM, Paton N, Winston A, Marcelin AG, Elbirt D, Hill A, Hadacek MB. Efficacy of protease inhibitor monotherapy vs. triple therapy: meta-analysis of data from 2303 patients in 13 randomized trials. HIV Med. 2016 May;17(5):358-67. doi: 10.1111/hiv.12348. Epub 2015 Dec 28. PMID 26709605
- [Background] Tubiana R, Mandelbrot L, Le Chenadec J, Delmas S, Rouzioux C, Hirt D, Treluyer JM, Ekoukou D, Bui E, Chaix ML, Blanche S, Warszawski J; ANRS 135 PRIMEVA (Protease Inhibitor Monotherapy Evaluation) Study Group. Lopinavir/ritonavir monotherapy as a nucleoside analogue-sparing strategy to prevent HIV-1 mother-to-child transmission: the ANRS 135 PRIMEVA phase 2/3 randomized trial. Clin Infect Dis. 2013 Sep;57(6):891-902. doi: 10.1093/cid/cit390. Epub 2013 Jun 12. PMID 23766338
- [Background] Andre-Schmutz I, Dal-Cortivo L, Six E, Kaltenbach S, Cocchiarella F, Le Chenadec J, Cagnard N, Cordier AG, Benachi A, Mandelbrot L, Azria E, Bouallag N, Luce S, Ternaux B, Reimann C, Revy P, Radford-Weiss I, Leschi C, Recchia A, Mavilio F, Cavazzana M, Blanche S. Genotoxic signature in cord blood cells of newborns exposed in utero to a Zidovudine-based antiretroviral combination. J Infect Dis. 2013 Jul 15;208(2):235-43. doi: 10.1093/infdis/jit149. Epub 2013 Apr 4. PMID 23559464
- [Background] Hleyhel M, Goujon S, Delteil C, Vasiljevic A, Luzi S, Stephan JL, Reliquet V, Jannier S, Tubiana R, Dollfus C, Faye A, Mandelbrot L, Clavel J, Warszawski J, Blanche S; ANRS French Perinatal Cohort Study Group. Risk of cancer in children exposed to didanosine in utero. AIDS. 2016 May 15;30(8):1245-56. doi: 10.1097/QAD.0000000000001051. PMID 26854809
- [Background] Mandelbrot L, Tubiana R, Le Chenadec J, Dollfus C, Faye A, Pannier E, Matheron S, Khuong MA, Garrait V, Reliquet V, Devidas A, Berrebi A, Allisy C, Elleau C, Arvieux C, Rouzioux C, Warszawski J, Blanche S; ANRS-EPF Study Group. No perinatal HIV-1 transmission from women with effective antiretroviral therapy starting before conception. Clin Infect Dis. 2015 Dec 1;61(11):1715-25. doi: 10.1093/cid/civ578. Epub 2015 Jul 21. PMID 26197844
- [Background] Valantin MA, Lambert-Niclot S, Flandre P, Morand-Joubert L, Cabie A, Meynard JL, Ponscarme D, Ajana F, Slama L, Curjol A, Cuzin L, Schneider L, Taburet AM, Marcelin AG, Katlama C; MONOI ANRS 136 Study Group. Long-term efficacy of darunavir/ritonavir monotherapy in patients with HIV-1 viral suppression: week 96 results from the MONOI ANRS 136 study. J Antimicrob Chemother. 2012 Mar;67(3):691-5. doi: 10.1093/jac/dkr504. Epub 2011 Dec 7. PMID 22160145
- [Background] Lambert-Niclot S, Flandre P, Valantin MA, Soulie C, Fourati S, Wirden M, Sayon S, Pakianather S, Bocket L, Masquelier B, Dos Santos G, Katlama C, Calvez V, Marcelin AG. Similar evolution of cellular HIV-1 DNA level in darunavir/ritonavir monotherapy versus triple therapy in MONOI-ANRS136 trial over 96 weeks. PLoS One. 2012;7(7):e41390. doi: 10.1371/journal.pone.0041390. Epub 2012 Jul 25. PMID 22848481